CLINICAL TRIAL: NCT03407027
Title: Evaluation of Triamcinolone's Efficacy on the Ultrasound- Guided Infiltration in the Quadratus Lumborum Syndrome: a Double Blind, Randomized, Controlled Study
Brief Title: Efficacy of Corticoid Infiltration in Quadratus Lumborum Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Braga (Other)
Collaborators: University of Minho (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CESHB 019/2016
Record Dates: First submitted 2017-10-12; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Low Back Pain
Keywords: Quadratus lumborum syndrome; ultrasound- guided infiltration
MeSH Terms: conditions — Low Back Pain | interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: In this randomized, double-blind trial, patients will be randomized into one of three groups. First group, infiltration of the quadratus lumborum muscle and fascia (with 40mg of triamcinolone and 10ml of levobupivacaine 0,25%). Second group, gluteus maximus and fascia infiltration with 40mg of triamcinolone and 10ml of levobupivacaine 0,25%. The last group, namely the control group, infiltration of the quadratus lumborum muscle and fascia with 10ml of levobupivacaine 0,25%.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadratus triamcinolone (Experimental): Quadratus lumborum muscle and fascia infiltration with 40mg of triamcinolone and 10ml of levobupivacaine 0,25%.
  Interventions: Drug: Quadratus triamcinolone
- Gluteus triamcinolone (Experimental): Gluteus maximus and fascia infiltration with 40mg of triamcinolone and 10ml of levobupivacaine 0,25%.
  Interventions: Drug: Gluteus triamcinolone
- Quadratus without triamcinolone (Active Comparator): Quadratus lumborum muscle and fascia infiltration with 10ml of levobupivacaine 0,25%.
  Interventions: Drug: quadratus without triamcinolone.

INTERVENTIONS:
Drug: Quadratus triamcinolone — 40mg of triamcinolone and 10ml of levobupivacaine 0,25%.
  Other Names: Quadratus lumborum infiltration with triamcinolone.
  Arms: Quadratus triamcinolone
Drug: Gluteus triamcinolone — 40mg of triamcinolone and 10ml of levobupivacaine 0,25%.
  Other Names: gluteus maximus infiltration with triamcinolone.
  Arms: Gluteus triamcinolone
Drug: quadratus without triamcinolone. — 10ml of levobupivacaine 0,25%.
  Other Names: quadratus lumborum infiltration without triamcinolone.
  Arms: Quadratus without triamcinolone

SUMMARY:
This study has the primary goal of evaluating the efficacy of corticoid infiltration in the quadratus lumborum syndrome, aiming to determine if there are benefits with the use of corticosteroids and if they exist, if this improvement comes only from the systemic effects of corticosteroid administration.

DETAILED DESCRIPTION:
This study has the primary goal of evaluating triamcinolone's efficacy on the ultrasound- guided infiltration in the quadratus lumborum syndrome, aiming to determine if there are benefits with the use of corticosteroids and if they exist, if this improvement comes only from the systemic effects of corticosteroid administration.

It is an interventional study, double-blinded and randomized, in a sample of patients followed in the Chronic Pain Unit (Hospital of Braga, Portugal), proposed for ultrasound infiltration of the quadratus lumborum muscle.

The selection of the patients will take into account the inclusion and exclusion criteria, until reach the required sample size (66 patients). The confirmation of the inclusion criteria will be done by a physiatrist blind to randomization.

Different protocols will be randomly applied to patients after obtaining written informed consent.

The techniques will be performed by two anesthetists. The data will be obtained through questionnaires filled out on the day of the technique and in the course of 1, 3 and 6 months in chronic pain consultation and by telephone call 72 hours after the procedure. It will be a psychologist, blind to randomization, to fill the questionnaires.

Patients will be also evaluated in consultation, at the same time, the course of 1, 3 and 6 months.

After the data collection it will be performed a statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

I) patients followed in the Chronic Pain Unit proposed to have ultrasound- guided infiltration of the quadratus lumborum muscle.

II) written informed consent.

III) presence of 4 of the following clinical criteria evaluated by a physiatrist:

* pain below the 12th rib and 5 cm lateral to the transverse process of L1 during palpation, with referred pain to the iliac crest;
* pain on palpation of the trigger points in the quadratus lumborum muscle;
* exacerbation of the pain with with postural changes when lying down, walking, sitting and/or squatting;
* lumbar pain with muscle stretching;
* painful palpation of trigger points at the level of L4 vertebral body, 1 to 2 cm above the iliac crest.

Exclusion Criteria:

* rheumatologic disease;
* psychiatric disease;
* neurological disease;
* history of anticoagulation use;
* pregnant patients;
* uncontrolled diabetes mellitus;
* patients on corticosteroid therapy;
* allergy to the medication to be used;
* anterior realization of ultrasound techniques for low back pain ;
* anterior realization, of invasive techniques, less than 6 months, with administration of medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of intervention. | 3 months after intervention.
  Evaluation of pain score using numerical rating scale (NRS), represented 0 with no pain and 10 with the worst pain imaginable. It will be evaluated the actual, average and worst intensity of pain. Efficacy of the procedure will be defined as greater or equal to 30% pain relief lasting at least 3 months.

SECONDARY OUTCOMES:
Pain evaluation | 6 months after intervention.
  Evaluation of pain score using numerical rating scale (NRS), represented 0 with no pain and 10 with the worst pain imaginable. It will be evaluated the actual, average and worst intensity of pain.
Quality of life. | 6 months after intervention.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Psychological status. | 6 months after intervention.
  To assess the level of anxiety and depression it will be used the HADS scale (Hospital Anxiety and Depression Scale).
  The HADS anxiety and depression subscales each consist of 7 items, and each item is rated on a 4-point scale; potential scores for each subscale range from 0 to 21. Patients with scores ≥8 on each subscale are considered symptomatic with general anxiety or depressive symptoms.
Complications and adverse effects caused by the intervention. | 72 hours after intervention.
  It will be asked to the patients for any adverse effect or complication including pain, hematoma, allergic reaction, paresthesias and decreased muscle strength.
Opioid consumption. | 6 months after intervention.
  Opioid intake will be converted in morphine equivalence in mg.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Cunha, MD, Principal Investigator — Hospital of Braga, Braga, Minho, Portugal, 4710-243
Locations (1):
- Hospital of Braga, Braga, Minho, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cid J, De La Calle JL, Lopez E, Del Pozo C, Perucho A, Acedo MS, Bedmar D, Benito J, De Andres J, Diaz S, Garcia JA, Gomez-Caro L, Gracia A, Hernandez JM, Insausti J, Madariaga M, Monino P, Ruiz M, Uriarte E, Vidal A. A modified Delphi survey on the signs and symptoms of low back pain: indicators for an interventional management approach. Pain Pract. 2015 Jan;15(1):12-21. doi: 10.1111/papr.12135. Epub 2013 Dec 9. PMID 24314001
- [Background] McEwen BS, Kalia M. The role of corticosteroids and stress in chronic pain conditions. Metabolism. 2010 Oct;59 Suppl 1:S9-15. doi: 10.1016/j.metabol.2010.07.012. PMID 20837196
- [Background] Pinto-Ribeiro F, Moreira V, Pego JM, Leao P, Almeida A, Sousa N. Antinociception induced by chronic glucocorticoid treatment is correlated to local modulation of spinal neurotransmitter content. Mol Pain. 2009 Jul 24;5:41. doi: 10.1186/1744-8069-5-41. PMID 19630968
- [Background] Iglesias-Gonzalez JJ, Munoz-Garcia MT, Rodrigues-de-Souza DP, Alburquerque-Sendin F, Fernandez-de-Las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in patients with chronic nonspecific low back pain. Pain Med. 2013 Dec;14(12):1964-70. doi: 10.1111/pme.12224. Epub 2013 Aug 15. PMID 23947760
- [Background] De Andres J, Adsuara VM, Palmisani S, Villanueva V, Lopez-Alarcon MD. A double-blind, controlled, randomized trial to evaluate the efficacy of botulinum toxin for the treatment of lumbar myofascial pain in humans. Reg Anesth Pain Med. 2010 May-Jun;35(3):255-60. doi: 10.1097/AAP.0b013e3181d23241. PMID 20921836